CLINICAL TRIAL: NCT00111462
Title: A Randomized, Open-Label Study of Darbepoetin Alfa (Novel Erythropoiesis Stimulating Protein, NESP) Using Fixed and Weight-Based Dosing for the Treatment of Anemia in Subjects With Non-Myeloid Malignancies Receiving Multicycle Chemotherapy
Brief Title: Evaluating Treatment of Anemia in Subjects With Non-Myeloid MalignanciesReceiving Multicycle Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20010102
Record Dates: First submitted 2005-05-20; First posted 2005-05-23 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Anemia; Non-Myeloid Malignancies; Cancer
Keywords: non-myeloid malignancy; chemotherapy-induced anemia
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa

SUMMARY:
The purpose of this study is to compare the effect of darbepoetin alfa administered in a weight based versus fixed dosing for the treatment of anemia in subjects with non-myeloid malignancies receiving multicycle chemotherapy.

ELIGIBILITY:
Inclusion Criteria: - Planned chemotherapy treatment - Anemia (hemoglobin concentration less than or equal to 11.0 g/dL) - Adequate renal and liver function - Eastern Cooperative Oncology Group (ECOG) 0 to 2 - Subjects must provide written informed consent Exclusion Criteria: - Known history of seizure disorder - Known primary hematologic disorder causing anemia other than non-myeloid malignancies - Unstable/uncontrolled cardiac condition - Clinically significant inflammatory disease - Known positive test for HIV infection - Transfusion within 4 weeks of randomization - Neutralizing antibodies to any erythropoietic agent - Treatment with erythropoietic therapy within 4 weeks before randomization - Received any investigational drug or device within 30 days before randomization - Pregnant or breast feeding - Not using adequate contraceptive precautions - Previously randomized into this study - Known hypersensitivity to any products to be administered - Concerns for subject's compliance

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
Achieving a hemoglobin concentration greater than or equal to 12.0 g/dL or a greater than or equal to 2.0-g/dL increase in hemoglobin concentration compared to baseline

SECONDARY OUTCOMES:
Time to and percentage of subjects with a hemoglobin response
Time to and percentage of subjects with hemoglobin correction
Hemoglobin concentration and change in hemoglobin concentration from baseline
Time to first RBC transfusion and percentage of subjects receiving a RBC transfusion

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Hesketh PJ, Arena F, Patel D, Austin M, D'Avirro P, Rossi G, Colowick A, Schwartzberg L, Bertoli LF, Cole JT, Demetri G, Dessypris E, Dobbs T, Eisenberg P, Fleischman R, Hall J, Hoffman PC, Laber DA, Leonard J, Lester EP, McCachren S, McMeekin S, Meza L, Miller DS, Nand S, Oliff I, Paroly W, Pawl L, Perez A, Raftopoulos H, Rigas J, Rowland K, Scullin DC Jr, Tezcan H, Waples J, Ward J, Yee LK. A randomized controlled trial of darbepoetin alfa administered as a fixed or weight-based dose using a front-loading schedule in patients with anemia who have nonmyeloid malignancies. Cancer. 2004 Feb 15;100(4):859-68. doi: 10.1002/cncr.11954. PMID 14770445
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com